CLINICAL TRIAL: NCT04528563
Title: Intravenous Ketorolac Vs. Morphine In Children Presenting With Suspected Appendicitis: A Pilot Single Center Non Inferiority Randomised Controlled Trial
Brief Title: Ketorolac for Moderate to Severe Abdominal Pain in Children
Acronym: KETO-APP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Mohamed Eltorki, MBChB, Assistant Professor, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 582125
Record Dates: First submitted 2020-08-23; First posted 2020-08-27 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Abdominal Pain; Appendicitis; Analgesia; Child, Only; Emergencies
MeSH Terms: conditions — Abdominal Pain; Appendicitis; Agnosia; Emergencies | interventions — Ketorolac Tromethamine; Morphine; Injections

STUDY DESIGN:
Intervention Model Description: double dummy design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketorolac Tromethamine (Experimental): IV ketorolac tromethamine, 0.5 mg/kg to a maximum of 30 mg plus IV morphine placebo;
  Interventions: Drug: Ketorolac Tromethamine 10 MG/ML
- Morphine Sulfate (Active Comparator): IV morphine 0.1 mg/kg to a maximum of 5 mg plus IV ketorolac placebo
  Interventions: Drug: Morphine Sulfate 10Mg/1mL Injection

INTERVENTIONS:
Drug: Ketorolac Tromethamine 10 MG/ML — Non-Steroidal-Anti-Inflammatory given intravenously.
  Arms: Ketorolac Tromethamine
Drug: Morphine Sulfate 10Mg/1mL Injection — Opioid commonly used for acute abdominal pain given intravenously.
  Arms: Morphine Sulfate

SUMMARY:
In children and adolescents (older than 6 years in age) who arrive in the pediatric emergency department because they have been having 5 days or less of abdominal pain (possible appendicitis), will patients who are treated with ketorolac get just as much pain relief as those patients treated with morphine?

To answer this research question, we will need a large number of patients in a study. To ensure we have enough patients, we must include many hospitals in different cities and provinces in the same study. Before doing this, though, we must first test a smaller version of the study in our center at McMaster Children's hosptial. The goal of doing this at McMaster first is to make sure or understand:

1. We can enroll enough people in our study over 1 year
2. We can make sure that all the information we collect from patients is complete and nothing is missing
3. Reasons behind why people don't want to participate in the study
4. How satisfied patients and their caregivers were with the study

DETAILED DESCRIPTION:
Background/Rationale: Appendicitis is the most common emergent surgical diagnosis among children between 5-17 years in age and accounts for 8000 admissions annually. Diagnosing appendicitis is time consuming (4-6 hours) as it requires laboratory tests and ultrasonography. This occurs while patients experience significant abdominal pain secondary to infection and localized or generalized peritonitis. Opioids have been the most prescribed analgesic for patients with suspected appendicitis, despite an ongoing opioid crisis. Our research shows that 60% of physicians use morphine or other opioids, while 40% will use non-steroidal anti-inflammatory drug (NSAID) or other non-opioids. Even though ketorolac (NSAID) is commonly used in the Emergency Department (ED) for renal colic, abdominal pain and migraine headaches, and has a safer side effect profile than morphine, all such uses in children are "off label" as there are virtually no controlled trials for children to inform practice.

Objective: To determine if it is feasible to conduct a large multi-centre randomized non inferiority trial comparing ketorolac to morphine for treating moderate to severe abdominal pain, in children 6 years in age or older, with clinically suspected appendicitis.

Hypothesis: We hypothesize that it will be feasible to conduct a large trial based on a recruitment rate of ≥40% of eligible patients approached for consent.

Study Design: Our trial is a single-centre, block randomized, non-inferiority, double-dummy, doubleblind, feasibility pilot trial. Patients ≥ 6 years in age, who have ≤ 5 days of moderate-severe pain as defined by our validated 11-point verbal numeric rating scale (VNRS) ≥ 5 and are being investigated for suspected appendicitis with intravenous (IV) access in situ or ordered, will be randomized to either: (1) IV ketorolac 0.5 mg/kg up to 30 mg (intervention) + IV morphine placebo, or (2) IV morphine 0.1 mg/kg up to 5 mg (active control) + IV ketorolac placebo. The total sample size is 100 participants. The study drugs will be identical in appearance, consistency and smell. The double-dummy design will ensure blinding is maintained for bedside clinical staff, research personnel and patients. Our study prioritized patient comfort and will largely mimic standard care. Pharmacologic co-interventions will be allowed but limited to acetaminophen (commonly used as first-line therapy). Participants in both groups will be allowed rescue therapy (morphine 0.5 mg/kg) within 60 minutes of our intervention. We will screen the ED daily for eligible patients as well as include all eligible patients for the New Investigator Fund (NIF)-funded quality improvement pathway we employed to streamline care for all ED appendicitis patients. We have a robust research program in the ED that includes students, a full-time research coordinator and several paid research assistants who screen eligible patients and approach them for consent and enrollment. Our entire project can be completed with NIF support within an 18-month study period.

Primary Outcome: Feasibility of our study design is the primary outcome of this pilot trial. Primary feasibility outcomes include: (1) proportion of patients consented from total eligible patients approached; (2) proportion of patients who completed clinical outcome assessment; and, (3) proportion of missing items on individual data collection forms. Our feasibility threshold is to recruit at least 40% of eligible patients who were approached to consent. Other thresholds include recruiting ≥8 participants/month on average and having at least 90% of participants complete all the outcome assessments at 30, 60, 90 and 120 minutes.

Summary: Acute pain in children and youth is an area that is understudied and affects thousands of Canadian children. Despite short -and long-term adverse effects including dependence, and well designed comparative effectiveness trials, opioids continue to be overused in surgical patients. Ketorolac is a promising well-established NSAID that is available for IV, has a better short-term side effect profile and is not known as a substance of misuse. Our pilot will provide valuable feasibility data for a larger, future multicenter trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6.0 years to <18 years: Children aged < 6 years of age at low risk for appendicitis and often present atypically.46,47
2. Duration of abdominal pain ≤ 5 days: Children with longer durations of acute abdominal pain are less likely to have appendicitis.18,48
3. A clinical decision to investigate for appendicitis as a possible etiology by the ED MD or RN. The physician or bedside nurse are suspicious of a diagnosis of appendicitis as a cause for the abdominal pain as reflected by the initiation of the appendicitis medical directive (an advanced nursing directive that allows nurses to order tests for patients with suspected appendicitis) and order laboratory tests and/or advanced imaging or directly consult pediatric surgery to rule out appendicitis.
4. Patient has an IV cannula in situ or ordered to be placed: we will not include patients without an IV ordered or established in order to ensure the study intervention is limited to the study drugs and is not associated with the performance of any invasive procedures.
5. Currently experiencing moderate to severe pain: self-reported pain score ≥5 using the VNRS at the time of enrollment.

Exclusion Criteria:

1. Previous enrollment in trial (to ensure all observations are independent and not paired)
2. NSAID use within 3 hours and/or opioid use within 2 hours prior to recruitment to avoid over-dosing and confounding
3. Caregiver and/or child cognitive impairment precluding the ability to self-report pain or respond to study questions
4. Chronic pain requiring daily analgesic use for other indications (e.g. naproxen for juvenile idiopathic arthritis): confounding
5. History of gastrointestinal bleeding, peptic or duodenal ulcer disease or inflammatory bowel disease, coagulation disorders, prior cerebrovascular bleeding, known arterio-vascular malformations: Bleeding risk
6. History of chronic and active renal disease, excluding renal calculi and urinary tract infections
7. History of chronic and active hepatocellular disease (excludes biliary stones, cholangitis or biliary duct pathology), as ketorolac is metabolized in the liver.
8. Known pregnancy at the time of enrollment, a positive pregnancy test in females ≥ 12 years in age or breastfeeding females due to the risk of premature closure of patent ductus arteriosus
9. Known hypersensitivity to NSAIDs or opioids (e.g. naproxen, ibuprofen, acetylsalicylic acid, ketoprofen or ketorolac, morphine, hydromorphone, fentanyl)
10. Absence of a parent/guardian for children who are < 16 years in age: youths who are ≥16 years can provide us with informed consent without the permission of a guardian
11. Inability to obtain consent due to a significant language barrier, in the absence of a native language translator

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-02-05 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Feasibility Outcomes | 2 hours
  proportion of patients consented from total eligible patients approached
Feasibility Outcomes | 2 hours
  Proportion of participants who completed outcome assessment at all time points
Feasibility Outcomes | 14 days
  Proportion of missing items on individual data collection forms (screening forms, baseline characteristics, outcome assessment, follow up survey)

SECONDARY OUTCOMES:
Study Satisfaction | 14 days
  Proportion of participants and caregivers who were satisfied with study procedures and interventions, on an 0-11 numeric satisfaction survey
Declining consent | 2 hours
  percentage and reasons for declining consent
withdrawing consent | 2 hours
  proportion of patients who withdrew consent
full study completion | 14 days
  proportion of patients who fully completed the study (baseline characteristics, outcome assessment and follow-up survey).

OTHER OUTCOMES:
Clinical Outcomes | 2 hours
  Within-group mean and standard deviation differences in pain as measured on verbal numerical pain scale (VNRS) for ketorolac and morphine at 30, 60, 90 and 120 minutes
Clinical Outcomes | 2 hours
  Proportion of participants who change their baseline pain category (mild 1 to 3, moderate 4 to 6, severe ≥7 on VNRS)
Clinical Outcomes | 2 hours
  Proportion of participants who achieved their desired pain state as determine on a numeric satisfaction scale (0-10)
Clinical Outcomes | 2 hours
  Time to effective analgesia (VNRS <3)
Clinical Outcomes | 6 hours
  Proportion of participants requiring rescue analgesia in each trial arm and the total amount administered as measured by morphine equivalent mg/kg within 6 hours of intervention
Clinical Outcomes | 14 days
  Frequency of missed appendicitis (diagnosed on a return visit within 7 days)
Clinical Outcomes | 24 hours
  Proportion of patients who had complete visualization of the appendix on ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Eltorki, MBChB, Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data and study-related documents will be available when the database has been locked and data has been unblinded.
Access Criteria: The data that support the findings of this study are available from the corresponding author (M.E), upon reasonable request

REFERENCES:
- [Derived] Eltorki M, Busse JW, Freedman SB, Thompson G, Beattie K, Serbanescu C, Carciumaru R, Thabane L, Ali S. Intravenous ketorolac versus morphine in children presenting with suspected appendicitis: a pilot single-centre non-inferiority randomised controlled trial. BMJ Open. 2022 Apr 5;12(4):e056499. doi: 10.1136/bmjopen-2021-056499. PMID 35383071